CLINICAL TRIAL: NCT03113435
Title: Patient Management During Major Abdominal Surgery: the Impact of a Hemodynamic Approach Oriented to Oxygen Consumption Optimization Compared to Standard Approach Targeting Preload-dependency and a Clinically-guided Strategy
Brief Title: Patient Management During Major Abdominal Surgery: an Oxygen Consumption Protocol Compared to Standard Approach
Acronym: HEART-CORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Flavia Torrini (Unknown); Alessandra Bisanti (Unknown); Eleonora Filipponi (Unknown); Domenica Luca Grieco (Unknown); Massimo Antonelli (Unknown); Liliana Sollazzi (Unknown); Valter Perilli (Unknown); Andrea Russo (Unknown); Pierpaolo Ciocchetti (Unknown)
Responsible Party: Principal Investigator, Antonio Maria Dell'Anna, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1305
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hemodynamic Instability
Keywords: CO2 gap; oxygen consumption; Stroke volume optimization

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard (No Intervention): In this group standard care will be provided to patients undergoing major abdominal surgery, regarding hemodynamic optimization
- NICE group (Active Comparator): In this arm patients will be treated according to stroke volume optimization described in NICE program
  Interventions: Other: Oxygen consumption optimization
- Oxygen consumption group (Experimental): In this arm patients will receive hemodynamic optimization based on their oxygen consumption need
  Interventions: Other: Oxygen consumption optimization

INTERVENTIONS:
Other: Oxygen consumption optimization — hemodynamic stability will be achieved through exploration of oxygen consumption need of the patient based on CO2gap/CaO2-CvO2 ratio
  Arms: NICE group; Oxygen consumption group

SUMMARY:
This study compares the actual standard of care with a new protocol to guide hemodynamic optimization during major abdominal surgery, which is more tailored on patient real needs. During general anesthesia metabolic needs of the body are markedly reduced and increase in CO may not be necessary. In addition, excessive fluid administration has been related to worse post-operative outcomes. We divide patients into three groups: the standard treatment group, the NICE protocol group and the intervention group. In this group we use the v-aCO2/CaO2-CvO2 as marker of tissue ability to increase their oxygen consumption in response to increased O2 delivery, and based on this index the administration of fluid. The principal aim is to optimize functional hemodynamics in order to reduce the fluid balance at the end of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients aged > 18 years
* acquisition of written informed consent
* Major abdominal surgery (major gastrointestinal surgery: DCP, gastrectomy, Miles, emicolectomy; gynecologic surgery: oncologic surgery) Surgery times ≥ 3 hours

Exclusion Criteria:

* Absolute contraindication to CVC placement
* pregnant women
* hepatic surgery
* laparoscopic surgery
* Major vascular surgery
* Dialysis treatment and kidney transplant surgery
* Severe heart failure (EF ≤ 35%)
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative fluid balance | surgery
  Perioperative fluid balance

SECONDARY OUTCOMES:
Survival at 28 days | 28 days after surgery
  Patients who survived at 28 days
Survival at hospital discharge | 1 day (Hospital discharge)
  Patient who survived at hospital discharge
Post-operative complication | 1 day (Hospital discharge)
  Increase in TnI, need for mechanical ventilation, infection, ICU admission, anastomotic leak, bleeding, AKI

CONTACTS AND LOCATIONS:
Overall Officials: Antonio M Dell'Anna, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli
Locations (1):
- Fondazione Policlinico A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided